CLINICAL TRIAL: NCT02668055
Title: Slow-release Tb4 Collagen and Chitosan Porous Sponge Scaffolds Skin Substitutes Treatment of Difficult to Heal Wounds Single-center Randomized Parallel Controlled Clinical Studies
Brief Title: Slow-release Tb4 Collagen and Chitosan Porous Sponge Scaffolds Skin Substitute Treatment is Difficult to Heal Wounds
Acronym: TB4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Academician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-005
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Wounds
Keywords: TB4; Difficult to heal
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TB4 (Experimental): Computing area was in proportion to the slow-release Tb4 collagen and chitosan porous sponge scaffolds skin substitute cells in wound, stick with wound edge skin suture, with vaseline gauze bandaging, controlled side not adding slow-release Tb4 collagen and chitosan porous sponge scaffolds skin substitutes
  Interventions: Biological: TB4

INTERVENTIONS:
Biological: TB4 — Computing area was in proportion to the slow-release Tb4 collagen and chitosan porous sponge scaffolds skin substitute cells stick in the wound surface

SUMMARY:
Evaluation of slow-release Tb4 collagen and chitosan porous sponge scaffolds skin substitutes the effectiveness of clinical trials for the treatment of difficult to heal wounds and security.

ELIGIBILITY:
Inclusion Criteria:

1. Meet difficult had 1 month or more to heal the wound patients
2. Who signed the informed consent of men or women older than 17 (pregnancy)
3. Has the ability to care for, has the ability to self signed informed consent, 7 to 17 years old must be signed by the guardian informed consent
4. The process of mental stability, can finish the test

Exclusion Criteria:

1. Known allergic to bovine collagen or gao min physique
2. the wound is greater than the10cm×10cm
3. People with mental illness, drug abusers and or other items
4. Pregnant women,Prepare a pregnancy or breast feeding women 5.3 months participated in other similar experiment

6.Serious infectious disease not controller 7.With surgery, such as severe trauma stress situation 8.Can not meet the requirement of the long-term follow-up of patients

Ages: 17 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months
  Tb4 collagen- chitosan porous sponge scaffolds skin substitute rate of wound healing, and healing

SECONDARY OUTCOMES:
Relative Wound Area Regression of 40% of More at 6 Week | 6week
  Subsistence the wound tissue(4 mm ×4 mm) biopsy samples, to determine the wound repair

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing Fu, Principal Investigator — Chinee PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China